CLINICAL TRIAL: NCT02218125
Title: A Phase I Study of Modified Vaccinia Ankara With Mosaic HIV Inserts in Healthy, HIV-Uninfected Adults, Some of Whom Have Previously Received an Adenovirus Type 26 ENVA.01 Vaccine
Brief Title: A Phase I Study of an HIV Vaccine in Healthy, HIV Uninfected Adults
Acronym: MENSCH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Crucell Holland BV (Industry)
Collaborators: US Military HIV Research Program (Network); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CR100965; IPCAVD006 (Other: Ragon Institute, Division of AIDS); HIV-V-A002 (Other: Crucell Holland BV)
Record Dates: First submitted 2014-08-14; First posted 2014-08-15 (Estimated); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Healthy
Keywords: Healthy; Human immunodeficiency virus type 1 (HIV-1) infection; Acquired immunodeficiency syndrome (AIDS); recombinant adenovirus (rAd) vector-based vaccines; Vaccination; Ad26.ENVA.01; Recombinant; Modified Vaccinia Ankara (MVA) vector-based vaccines
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Infections; Dyschromatosis symmetrica hereditaria 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (4):
- Group 1- MVA Mosaic (Experimental): Healthy volunteers not previously vaccinated with Ad26.ENVA.01 will be administered Modified Vaccinia Ankara (MVA) Mosaic at Week 0 and at Week 12.
  Interventions: Biological: MVA Mosaic
- Group 2 - Placebo (Placebo Comparator): Healthy volunteers not previously vaccinated with Ad26.ENVA.01 will be administered placebo at Week 0 and at Week 12.
  Interventions: Biological: Placebo
- Group 3 - MVA Mosaic (Experimental): Healthy volunteers previously vaccinated with Ad26.ENVA.01 will be administered MVA Mosaic at Week 0 and at Week 12.
  Interventions: Biological: MVA Mosaic
- Group 4- Placebo (Placebo Comparator): Participants previously vaccinated with Ad26.ENVA.01 will be administered placebo at Week 0 and at Week 12.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: MVA Mosaic — 0.5 mL (1x10E8 pfu) MVA Mosaic (comprised of MVA Mosaic 1 and MVA Mosaic 2 mixed in a 1:1 ratio before administration) will be administered by intramuscular (IM) injection.
  Arms: Group 1- MVA Mosaic; Group 3 - MVA Mosaic
Biological: Placebo — 0.5 mL Sodium Chloride Injection USP, 0.9%will be administered by intramuscular (IM) injection.
  Arms: Group 2 - Placebo; Group 4- Placebo

SUMMARY:
The purpose of this study is to assess the safety and tolerability of Modified Vaccinia Ankara (MVA) Mosaic vaccine in healthy adult participants.

DETAILED DESCRIPTION:
This is a Phase I, placebo-controlled (the use of an inactive substance identical in appearance to the active vaccine), double-blind (neither the participant or study personnel will know the identity of the treatment administered) study where participants will be randomized (treatment type assigned by chance) to receive a Modified Vaccinia Ankara (MVA) Mosaic vaccine (at 1x10E8 pfu) or placebo. This design is intended to reduce the likelihood of observer and selection bias, provide control for confounding variables, and aid an unbiased analysis of the study results. The study will include 4 groups of participants, 2 groups having previously been vaccinated with Ad26.ENVA.01 (A recombinant adenovirus [rAd] vaccine for HIV-1) and 2 groups not previously vaccinated with Ad26.ENVA.01. Participants will be randomized in a 4:1 ratio to receive either a MVA Mosaic vaccine or placebo. The trial comprises a 4-week screening period, a 12-week vaccination period during which participants will be vaccinated at baseline (Day 1) and Week 12 (Day 84), and a 40-week follow-up period to the final visit at Week 52.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults (determined by medical history, physical examination, and clinical judgment)
* HIV uninfected
* Female participants of child bearing potential must have a negative serum β-human chorionic gonadotrophin pregnancy test at the screening visit and immediately prior to each vaccine/placebo administration, practice adequate birth control measures from 28 days prior to the first vaccine/placebo administration through to at least 3 months after the final vaccine/placebo administration
* Male participants who are sexually active with a woman of childbearing potential and has not had a vasectomy must agree to use a double barrier method of birth control, e.g. either condom with spermicidal foam/gel/film/cream/suppository or partner with occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository

Exclusion Criteria:

* Confirmed HIV-1/-2 infection
* Chronic active hepatitis B or hepatitis C or active syphilis infection. Active syphilis documented by exam or serology unless positive serology is due to past treated infection
* Within the 12 months prior to enrollment: a history of newly acquired syphilis, gonorrhea, non-gonococcal urethritis, herpes simplex virus type 2 (HSV2), Chlamydia, pelvic inflammatory disease (PID), trichomonas, mucopurulent cervicitis, epididymitis, proctitis, lymphogranulomavenereum, chancroid, or hepatitis B
* A woman who is breastfeeding
* Any clinically significant acute or chronic medical condition that, in the opinion of the investigator, would preclude participation
* Major surgery within the 4 weeks prior to study entry or planned major surgery through the course of the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2014-09-23 (Actual); Primary Completion 2015-11-30 (Actual); Study Completion 2015-11-30 (Actual)

PRIMARY OUTCOMES:
The Number of Participants who Experience Adverse Events Within 28 days After Vaccination | For 28 days following vaccination on Day 1 and Day 84
  In addition to the number of participants who experience adverse events within the time frame of 28 days after each vaccination, all adverse events that occur from the signing of the informed consent through to the last study visit (Visit 10 [Day 365]) will be reported.
The Number of Participants who Experience Reactogenicity Symptoms Following Vaccination | 1 week following vaccination on Day 1 and Day 84
  Reactogenicity symptoms monitored following vaccination will include erythema (redness), induration (hardening), and local pain/tenderness, itching, swelling, or warmth at the site of injection, temperature (fever >37.7 degree Celsius); fatigue (extreme tiredness), headache, myalgia (muscle pain), arthralgia (joint pain), chills, nausea, vomiting, rashes, and itching (general and local)

SECONDARY OUTCOMES:
The Number of Participants With Humoral Immune Responses | 4 weeks after the second vaccination
  Humoral immune responses will be evaluated by the detection of env-specific binding antibody.
Durability of Immune Response | 6, 9, and 12 months after the first vaccination
  Determined by humoral immune response assays.
The Number of Participants With T-cell Responses Following Vaccination | 4 weeks after the second vaccination
  T-cell responses to be determined by epitope mapping.

CONTACTS AND LOCATIONS:
Overall Officials: Crucell Holland BV Clinical Trial, Study Director — Crucell Holland BV
Locations (1):
- Boston, Massachusetts, United States

REFERENCES:
- [Derived] Baden LR, Walsh SR, Seaman MS, Cohen YZ, Johnson JA, Licona JH, Filter RD, Kleinjan JA, Gothing JA, Jennings J, Peter L, Nkolola J, Abbink P, Borducchi EN, Kirilova M, Stephenson KE, Pegu P, Eller MA, Trinh HV, Rao M, Ake JA, Sarnecki M, Nijs S, Callewaert K, Schuitemaker H, Hendriks J, Pau MG, Tomaka F, Korber BT, Alter G, Dolin R, Earl PL, Moss B, Michael NL, Robb ML, Barouch DH; IPCAVD006/RV380/HIV-V-A002 Study Group. First-in-Human Randomized, Controlled Trial of Mosaic HIV-1 Immunogens Delivered via a Modified Vaccinia Ankara Vector. J Infect Dis. 2018 Jul 13;218(4):633-644. doi: 10.1093/infdis/jiy212. PMID 29669026